CLINICAL TRIAL: NCT02910999
Title: A National, Prospective, Non-Interventional Study (NIS) of Nivolumab (BMS-936558) In Patients With Locally Advanced Or Metastatic Non-Small Cell Lung Cancer (NSCLC) With Squamous and Non-Squamous Histology (Stage IIIB/IV) After Prior Chemotherapy
Brief Title: Real-Life Study With Nivolumab (BMS-936558) in Advanced NSCLC Patients After Prior Chemotherapy
Acronym: ENLARGE-Lung
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-580
Record Dates: First submitted 2016-09-02; First posted 2016-09-22 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NSCLC patients with squamous tumor histology
- NSCLC patients with non-squamous tumor histology

SUMMARY:
This study intends to describe the real-life effectiveness and safety of nivolumab in advanced NSCLC patients in Germany, as well as the patient profile, pattern of use and the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of locally advanced or metastatic NSCLC, Stage IIIB/Stage IV
* Decision to initiate a treatment with Nivolumab for the first time already undertaken by physician
* Males and Females, ≥18 years of age

Exclusion Criteria:

* Current primary diagnosis of a cancer other than advanced NSCLC. Example: A cancer other than NSCLC that requires systemic or other treatment.
* Pre-treatment with Nivolumab and/or Ipilimumab (pre-treatment with checkpoint-inhibitors other than Nivolumab and Ipilimumab, and Tyrosine Kinase Inhibitors(TKIs) is allowed)
* Current participation in an interventional clinical trial for treatment of NSCLC. (Patients who have completed their participation in an interventional trial or who are not receiving study drug anymore and who are only followed-up for overall survival can be enrolled. For blinded studies, the treatment administered needs to be known)

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both cohorts will be recruited in different sites. Office-based as well as outpatient units in clinics.
Sampling Method: Probability Sample
Enrollment: 868 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Approximately 5 years

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Approximately 5 years
Overall Response Rate (ORR) | Approximately 5 years
Best Overall Response Rate (BORR) | Approximately 5 years
Best Overall Response (BOR) | Approximately 5 years
Duration of Response (DOR) | Approximately 5 years
Distribution of socio-demographic characteristics in adult patients diagnosed with advanced NSCLC | At baseline and for up to 5 years
Distribution of clinical characteristics in adult patients diagnosed with advanced NSCLC | At baseline and for up to 5 years
Distribution of treatment patterns in adult patients diagnosed with advanced NSCLC | At baseline and for up to 5 years
Distribution of Incidence of All Adverse Events (AEs) | Approximately 5 years
Distribution of Severity of All Adverse Events (AEs) | Approximately 5 years
Distribution of Management of All Adverse Events (AEs) | Approximately 5 years
European Quality of Life-5 Dimensions (EQ-5D) | At baseline and for up to 5 years
Lung Cancer Symptom Scale (LCSS) | At baseline and for up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Frankfurt, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html